CLINICAL TRIAL: NCT06284031
Title: Cervical Cancer Brachytherapy With Interstitial Needles in 3 Fractions: Dosimetric and Clinical Outcomes
Brief Title: Cervical Cancer Brachytherapy With Interstitial Needles in 3 Fractions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Brachy Study
Record Dates: First submitted 2023-07-25; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-08

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3 fractions (Experimental)
  Interventions: Procedure: 3 fractions HDR brachytherapy

INTERVENTIONS:
Procedure: 3 fractions HDR brachytherapy — The 3 fractions of HDR brachytherapy may be delivered in the following ways:
  Option 1: 3 insertions over 2 non-consecutive days:
  Option 2: 3 insertions over 3 non-consecutive days

SUMMARY:
Aim To determine the feasibility and safety of 3 fractions of high dose rate (HDR) brachytherapy with interstitial needles for cervical cancer in the outpatient setting

Primary objective To determine the clinical outcome (2-yr local control rate, loco-regional control rate, progression free survival and overall survival)

Secondary objective To determine the long-term toxicities of this regimen based on CTCAE v5

DETAILED DESCRIPTION:
This study is designed as a single arm phase II prospective study that will be open for recruitment for approximately 3 years. An estimated 56 cervical cancer patients treated in NUH will be recruited.

Pre-treatment Assessment

1. Case reviewed in gynae multidisciplinary meeting
2. Detailed gynaecologic assessment on diagnosis
3. Staging scan - MRI pelvis, CT TAP or PET CT
4. Baseline blood result - Full blood count, renal panel, liver panel, coagulation profile and Group screen and match

Treatment

All patients will be registered and reviewed in NUH Radiotherapy Centre. Written consent will be obtained if patient is agreeable to be recruited.

Brachytherapy A pre-brachytherapy planning magnetic resonance imaging (MRI) scan is performed to evaluate the response and extent of the parametrial involvement if any, as well as to determine the ideal placement of interstitial needles to achieve optimal coverage. The applicator to be used should be chosen prior to BT if possible. Twenty-four hours prior to the procedure, oral fleet is given to the patient to ensure adequate bowel preparation.

The 3 fractions of HDR brachytherapy may be delivered in the following ways:

Option 1: 3 insertions over 2 non-consecutive days:

9 Gy to the HRCTV in the first fraction on day 1 of the brachytherapy procedure and 7 Gy x 2 fractions at least 6 hours apart on day 2, retaining the same brachytherapy applicators of the second insertion for the final fraction.

Option 2: 3 insertions over 3 non-consecutive days 8Gy to the HRCTV per fraction per day for 3 non-consecutive days. Acute and late radiation toxicities will be scored according to Common Terminology Criteria for Adverse Events (CTCAE), version 5 Patients will be followed up at 1 month with a physical examination and with an MRI of the cervix within 3 months post procedure.

Patients will subsequently be followed up every 3 monthly with vaginal examination for the next 2 years. At each follow-up, toxicity will be recorded as per the CTCAE.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years old and above
2. Histologically proven squamous cell carcinoma, adenocarcinoma, adenosquamous or poorly differentiated cervical cancer
3. Clinically or radiologically stage IB - IVA cervical cancer based on TNM 8th Edition
4. ECOG performance status 0, 1, or 2
5. To complete external beam radiotherapy and brachytherapy in NUH
6. Written, voluntary informed consent
7. Patients must be accessible for follow up and management in NUH

Exclusion Criteria:

1. Post operative cervical cancer cases
2. Pregnant or breastfeeding women

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As cervical cancer patients are females, we will only be recruiting female patients.
Enrollment: 56 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Local control rate | 2 years from time of recruitment
  Percentage of patients who recurred at the site of the initial primary (the cervix).
Loco-regional control rate | 2 years from time of recruitment
  Percentage of patients who recurred in the pelvis or regional lymph nodes (not in cervix).
Progression-free survival (PFS) | 2 years from time of recruitment
  Percentage of patients who develop first evidence of cancer recurrence.
Overall survival (OS) | 2 years from time of recruitment
  Percentage of patients who died from any cause

SECONDARY OUTCOMES:
Long term toxicities | 2 years from time of recruitment
  To determine the long-term toxicities of this regimen based on CTCAE v5

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Koh, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No